CLINICAL TRIAL: NCT06524791
Title: Evaluation of the Prevalence of Faecal Bacteriophage Carriage in Patients With Digestive Symptoms.
Brief Title: Prevalence of Faecal Bacteriophage in Patients With Digestive Symptoms
Acronym: PREPHAGE
Status: Not yet recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, HARTARD Cédric, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2023-0323
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Gastroenteritis
Keywords: bacteriophages
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — stool sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- immunocompetent: immunocompetent patients with digestive symptoms (n=150)
  Interventions: Other: bacteriophage detection
- immunocompromised: immunocompromised patients with digestive symptoms (n=150)
  Interventions: Other: bacteriophage detection

INTERVENTIONS:
Other: bacteriophage detection — bacteriophage detection

SUMMARY:
Define the prevalence of fecal phage carriage in individuals with digestive symptoms (i) Determine the concentrations of infectious fecal phages in the stools of individuals with digestive symptoms (detection by culture)

(ii) Determine fecal phage genome concentrations in the stools of individuals with digestive symptoms (PCR detection)

(iii) Explore factors that could impact fecal phage carriage (patients with digestive symptoms vs. healthy individuals, immunocompromised patients vs. immunocompetent patients)

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60.
* Persons having developed gastrointestinal symptoms justifying microbiological stool testing at the time of hospitalization.
* Person having received full information on the organization of the research and not having objected to the use of this data

Exclusion Criteria:

* Persons covered by articles L. 1121-5, L. 1121-7 and L1121-8 of the French Public Health Code.
* Pregnant or breast-feeding women,
* Minors (not emancipated),
* Adult subject to a legal protection measure (guardianship, curatorship, safeguard of justice),
* Persons of full age who are unable to give their consent.
* Persons deprived of their liberty by a judicial or administrative decision, persons under psychiatric care by virtue of articles L. 3212-1 and L. 3213-1.

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: patients hospitalized at the CHRU de Nancy with digestive symptoms requiring microbiological stool analysis
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
prevalence of faecal phage carriage | baseline
  define the prevalence of faecal phage (coliphage) carriage in individuals presenting with digestive symptoms.

SECONDARY OUTCOMES:
concentrations of infectious fecal phages | baseline
  Determine the concentrations of infectious fecal phages in the stools of individuals with digestive symptoms (detection by culture)
fecal phage genome concentrations | baseline
  determine fecal phage genome concentrations in the stools of individuals with digestive symptoms (PCR detection)

CONTACTS AND LOCATIONS:
Overall Officials: Cédric Hartard, Principal Investigator — CHRU Nancy
Locations (1):
- CHRU Nancy, Nancy, France